CLINICAL TRIAL: NCT06252727
Title: Fluorescent Aided Resection and Evaluation of Soft Tissue Sarcomas (FLARES)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI choice.
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2074423
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Soft Tissue Sarcoma; Soft Tissue Sarcoma Adult
MeSH Terms: conditions — Sarcoma | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aminolevulinic acid (5-ALA) (Experimental): 20 mg/kg body weight of 5-ALA orally at 3-4 hours prior to surgical resection. 5-ALA fluorescence will be used to evaluate the resected tumor per gross margins and identifying further areas of fluorescing tissues beyond the gross tumor margins.
  Interventions: Drug: Aminolevulinic Acid

INTERVENTIONS:
Drug: Aminolevulinic Acid — Given PO
  Other Names: 5-ALA; Gleolan

SUMMARY:
This will be a prospective pilot study that will evaluate 20 patients who were diagnosed with FNCLCC Grade 2 or 3 soft tissue sarcomas and will undergo surgical resection. Based upon the FDA label, successful protocols used for intraoperative fluorescence-guided visualization for glioma resections, and on drug company current dosing recommendation for this study, patients will be administered 20 mg/kg body weight of 5-ALA orally at 3-4 hours prior to surgery. The use of 5-ALA fluorescence will be relevant for evaluating the resected tumor per gross margins and identifying further areas of fluorescing tissues beyond the gross tumor margins.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE: I. Demonstrate the feasibility of 5-ALA-aided fluorescent visualization of STS versus surrounding tissues.

SECONDARY OBJECTIVE:

I. Demonstrate the efficacy of tumor and surgical margin resections by a gross and histological analysis of fluorescing and non-fluorescing samples immediately after removal.

II. Assess the safety profile of fluorescence-guided surgery (FGS) for STS utilizing 5-ALA.

OUTLINE: Patients will be administered 20 mg/kg body weight of 5-ALA orally at 3-4 hours prior to surgical resection. Intraoperative fluorescence-guided visualization will be used for evaluating the resected tumor per gross margins and identifying further areas of fluorescing tissues beyond the gross tumor margins.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of any subtype of primary Grades 2 or 3 soft tissue sarcomas (STS), per biopsy evaluation by a pathologist, according to Fédération Nationale des Centres de Lutte Contre le Cancer (FNCLCC).
* Treatment decision includes planned surgical resection of STS.
* Age ≥18 years at time of consent.
* ECOG Performance Status 0 - 1 (see Appendix)
* Hematology and blood chemistry parameters defined by:

  * Leukocytes ≥ 3 × 109/L
  * Absolute neutrophil count ≥ 1.5 × 109/L
  * Platelets ≥ 100 × 109/L, transfusions may be used to raise platelets to ≥ 100 × 109/L (no washout required)
  * Hemoglobin ≥ 9 g/dL, transfusions may be used to raise Hgb to ≥ 9 g/dL (no washout required)
  * Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
  * Aspartate transaminase (AST) / alanine transaminase (ALT) ≤ 2.5 × institutional ULN
  * Creatinine within normal institutional limits OR creatinine clearance ≥ 30 mL/min/1.73 m2 for patients with creatinine above institutional ULN
* Participants of reproductive potential must agree to using adequate contraception (e.g., hormonal or barrier method of birth control; abstinence, an intrauterine device) for the duration of study participation (including dosing interruptions) and up to 42 days after end of study intervention; or be surgically sterilized (e.g., hysterectomy, tubal ligation, or vasectomy).
* Ability to swallow study agent.
* Ability to understand and willingness to sign an informed consent form.
* Ability and stated willingness to adhere to the study visit schedule and other protocol procedures/requirements for the duration of the study.

Exclusion Criteria:

* Acute/chronic forms of porphyria.
* Uncontrolled, known concurrent illness, including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness.
* Patient has had chemotherapy, tumor resection, or radiation treatment ≤ 21 days prior to surgery.
* Simultaneous participation in another clinical trial ≤ 21 days of enrollment or during the duration of the study period.
* Planned use of other potentially phototoxic substances (e.g., St. John's wort, griseofulvin, thiazide diuretics, sulfonylureas, phenothiazines, sulfonamides, quinolones and tetracyclines), and topical preparations containing aminolevulinic acid (5-ALA) for 24 hours during the perioperative period (defined as 24 hours prior to surgery to up to 24 hours post surgery).
* Pregnant or planning to become pregnant during study participation or breastfeeding.
* Any condition that in the opinion of the investigator would prohibit the understanding or rendering of informed consent or interfere with the participant's safety or compliance while on trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of 5-ALA-aided fluorescent visualization of STS versus surrounding tissues | Up to 2 years
  Ability of 5-ALA to provide intraoperative fluorescent visualization of STS versus surrounding tissues as assessed by the fluorescence of the surgical bed and hemisected soft tissue sarcoma (STS) after resection. This will be assessed during the surgical procedure and recorded via imaging and videography to analyze fluorescent visualization

SECONDARY OUTCOMES:
Efficacy of tumor and surgical margin resections by a gross and histological analysis of fluorescing and non-fluorescing samples immediately after removal. | Up to 2 years
  Verification of margins and disease tissue by sarcoma pathologist.
Disease free survival. | Up to 2 years
  Time to development of recurrent disease or death from any cause.
Incidence of treatment related adverse events. | Up to 2 years
  Number of intervention-related adverse events (AEs) per NCI CTCAE v5.0 as assessed through patient reported outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Steven W Thorpe, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States